CLINICAL TRIAL: NCT07295171
Title: HELP Study - Towards High Throughput and Efficient Long-axial PET With Oral [18F]FDG
Acronym: HELP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: H25-02148
Record Dates: First submitted 2025-09-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Multiple Cancers; Multiple Indications Cancer; Feasibility Studies
Keywords: Oral FDG; LAFOV; Long-axial Field-of-view Scanner; Quadra; Low-dose Oral Radiopharmaceuticals

STUDY DESIGN:
Intervention Model Description: Step 1: N=5 Dosimetry (1h dynamic scan post ingestion of the radiopharmaceutical) and initial assessment of biodistribution at 2h Step 2: N=3 To determine if patients may leave the uptake room, move gently and consume water during the longer waiting period before the static scan. To determine if 3h post ingestion is sufficient.
  Step 2a: N=3-12 p.r.n. Interim step if further refinements to patient behavior or the uptake time is necessary. If not required, proceed to Step 3 Step 3: N=7 Assessment of final protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral FDG scan and standard of care FDG scan (Experimental): Participants will receive their standard of care FDG scan and then an Oral FDG scan within two weeks.
  The standard of care FDG scan will involve IV administration of FDG. The Oral FDG scan will involve FDG diluted in 50ml (approx.) of water to be consumed by mouth.
  The length of the oral FDG scans and its comparison to the standard FDG scan depends on which step the study is currently on. Please refer to the Study Design for details on the Oral FDG scan.
  Interventions: Diagnostic Test: Oral FDG scan

INTERVENTIONS:
Diagnostic Test: Oral FDG scan — Evaluating the feasibility, scan quality and ease of administration when FDG is consumed orally rather than administered by IV.

SUMMARY:
Typically, PET scans involve an IV injection of 18F-FDG that helps identify cancer. Patients are scanned 60 minutes after injecting 18F-FDG. This study aims to assess the feasibility of a different method of administration - oral ingestion (rather than IV) of 18F-FDG through delayed imaging to identify the optimal time for scanning after consuming the drug. The study will aim to recruit 15-24 individuals who will receive two PET scans - one using delayed oral 18F-FDG imaging and a second regular 18F-FDG. The analysis will focus on establishing a suitable protocol for this administration route while considering patient preference and image quality.

DETAILED DESCRIPTION:
Purpose:

Radiopharmaceutical:

18F-FDG is the most commonly PET radiopharmaceutical because of it's wide availability and its use across oncological indications. This tracer binds to the glucose molecules in the body to outline tumor cells. Typically it is administered through IV but this study will explore its feasibility when consumed orally.

Marketed device:

BC Cancer has recently acquired a Long Axis Field of View (LAFOV) machine (called Siemens Quadra) that can scan patients in 1-2 minutes rather than 20 minutes on a more commonly found SAFOV scanner. LAFOV scanners can provide much higher resolutions of scans compared to SAFOV.

The purpose of this study is to create an optimal protocol to scan patients with oral 18F-FDG on the LAFOV machine to utilize this machine's high resolution and fast throughput. From previous studies, investigators know that oral 18F-FDG is absorbed differently when compared to 18F-FDG through IV (Srinivas et al, 2020). To better inform the protocol, this study will use a delayed imaging method to assess the absorption during uptake time and image quality resulting from this different route of administration. Lastly, the study will compare scan results from oral 18F-FDG scans with that of regular 18F-FDG scans to assess the benefits and feasibility in a clinic setting.

Justification:

PET scans typically involve the injection of 18F-FDG through IV 60 minutes before the patient is scanned. The radiopharmaceutical is absorbed by the body during the uptake time of 60 minutes and the images resulting from the scan can be used to identify cancerous cells. This process requires the patient to be resting during uptake period to ensure the tracer isn't absorbed into muscles due to activity. Additionally, venous access could result in extravasation, bruises at injection site, patient discomfort and longer prep time for staff. In a clinic setting with higher throughput demands, number of uptake rooms and prep time are often the rate-limiting factor.

Consuming 18F-FDG orally results in a much slower uptake process (Srinivasan et al, 2020) and may eliminate the need to confine patients to a room during uptake. The LAFOV scanner is capable of scanning more patients in a period of time than uptake rooms are available. Therefore, not requiring patients to remain in a room may allow more patients to be scanned faster.

Research Design:

This study is a prospective, open-label, single-cohort, phase I study to determine the feasibility of scanning with oral FDG. Participation will involve one scan with regular FDG and one scan with oral FDG within 14 days of each other. The study will be divided into 3 steps to test different uptake times and patient activity levels for protocol optimization. Participants cannot participate in more than 1 step.

This small pilot study aims to determine the optimal examination protocol and feasibility of ambulatory and oral application of [18F]FDG in conjunction with a latest-generation high-sensitivity LAFOV scanner system. Comparisons between the oral and SOC intravenous scans will be made using descriptive statistics.

Sample size estimate:

The sample size for study will be a pragmatic determination based on feasibility considerations. So as not to unduly burden the study with the long 1h dosimetry requirements from kinetic scanning, the investigators shall perform dosimetry in 5 subjects.

The sample size is designed to afford a preliminary check of the protocol's feasibility before moving to the next stage. Once the final protocol is reached (Step 3) - a minimum of N=10 patients will be available with a comparable protocol for an initial estimate of the technique's performance.

The data generated will afford a power calculation for a phase II trial if appropriate STEP 1: N=5 STEP 2: N=3 STEP 2(a): N=3 (optional) STEP 3: N=7

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years
* Participants who have received a standard of care [18F]FDG PET/CT and are willing to undergo a study specific oral [18F]FDG PET/CT within 2 weeks.

Exclusion Criteria:

Participant Inclusion Criteria

* Age ≥19 years
* Participants who have received a standard of care [18F]FDG PET/CT and are willing to undergo a study specific oral [18F]FDG PET/CT within 2 weeks.

Participant Exclusion Criteria

* Pregnant or breast-feeding
* Medically unstable (e.g., acute illness, unstable vital signs)
* Urinary incontinence/catheter.
* Immobile, frail or vulnerable patients who cannot leave the department and would require an uptake room in any case.
* Patients whose fasting blood sugar at the SOC PET was >11.0 mmol/l
* Unable to swallow.
* Patients with nasogastric tubes, percutaneous gastrostomy or other non-anatomical routes for nutrition.
* Unable to lie flat for 1h (subset of participants - first 5 participants only).
* Claustrophobia requiring medication.
* Undergoing active treatment or assessment of an upper digestive tract tumor (stomach/esophagus)
* Unable to provide written consent
* Patients receiving biguanide anti-hyperglycemic agents (e.g. Metformin).
* Insulin dependent diabetics.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of hours for radiopharmaceutical to be cleared from stomach for optimal imaging | Periprocedural
  To identify an acceptable imaging time to achieve gastric clearance of the radiopharmaceutical (time post administration in hours)
Image quality compared to the standard of care FDG scan | within 2 weeks of the scan
  They shall be asked to rate the quality of each scan on a five point Likert scale (5 being the highest, 1 being the lowest).
To assess participant preference for this method of administering radiopharmaceutical | periprocedural
  Participants will be given a sheet with 4 questions to answer about their experiences with the new mode of administration. The questions are:
  1. Which scan did you prefer: oral or the injection? Why?
  2. Where do you prefer to wait: in the uptake room or outside the department? Why?
  3. What did you do during the waiting time for the study scan? (select all that apply) Walk / read/ listen to music / talk with friends/family / other (specify)
  4. Did you drink water while waiting? How much __ mL

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Vancouver, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No